CLINICAL TRIAL: NCT01151878
Title: Glucomannan in Treating Childhood Functional Constipation: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Glucomannan for Childhood Functional Constipation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB/127/2008
Record Dates: First submitted 2010-05-07; First posted 2010-06-29 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Functional Constipation
Keywords: constipation; children
MeSH Terms: conditions — Constipation | interventions — (1-6)-alpha-glucomannan; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and researchers conducting the study were blinded. Intervention products were prepared in sachets centrally by the hospital pharmacy by a person not involved in the conduct of the trial. The active product and placebo were packaged in identical sachets and labeled with one of two codes, each allocated to the experimental product or placebo. This procedure was performed by an independent pharmacist, who was the only person aware of the codes' meaning. The appearance and texture of the dry products were identical.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucomannan (Experimental): glucomannan preparation in sachets: 1 saschet of 1.26g 2 times per day (daily dosage 2,52g); duration of intervention: 4 weeks
  Interventions: Dietary Supplement: Glucomannan
- Placebo (Placebo Comparator): maltodextrin prepared in sachets (1,3 g per sachet); 2 sachets per day; duration of intervention: 4 weeks
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Glucomannan — 1.26 g per sachet; 2 sachets per day for 4 weeks.
  Other Names: Dicoman Junior, Vitis Pharma
  Arms: Glucomannan
Dietary Supplement: maltodextrin — prepared in sachets (1.3g); 2 sachets per day for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether administration of glucomannan (dietary fiber) is effective in treating functional constipation in children.

DETAILED DESCRIPTION:
Constipation is a common condition in children. In many patients symptoms persist to adulthood and decrease quality of life. The standard treatment, mostly osmotic laxatives such as lactulose or polyethyleneglycols, are often ineffective and may cause adverse events. Therefore, alternative treatment measures are being searched for.

Glucomannan, a water-soluble fiber polysaccharide from the tubers of the Japanese Konjac plant, has been reported to be effective in constipated children. To date, 2 randomized trials were performed.1,2 One evaluated the effect as glucomannan as an adjunct to standard treatment.1 Another was conducted in neurologically impaired children, who constitute a specific population that cannot be compared to patients with functional constipation.2 In both trials, the number of patients was relatively small.

Well-powered, randomized controlled study is required to evaluate clinical effectiveness of glucomannan as a sole treatment in childhood functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* functional constipation diagnosed according to Rome Criteria III (duration of symptoms for at least 2 months prior to study inclusion)
* age 3 to 16 years
* informed consent from parents and/or child

Exclusion Criteria:

* organic cause of defecation disorders (Hirschsprung's disease, spinal anomalies or anorectal pathology; history of gastro-intestinal surgery)
* mental retardation
* metabolic disease (e.g. hypothyroidism)
* irritable bowel syndrome
* intake of medications influencing gastrointestinal motility

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
treatment success | 1 week
  paasing at least 3 stools per week with no episodes of soiling

SECONDARY OUTCOMES:
stool frequency | 1 week
  number of stools passes per week
soiling | 1 weeks
  number of episodes of soiling per week
hard stools or painful defecations | 1 week
  number of hard stools passed or painful defecations per week
abdominal pain | 1 week
  number of episodes of abdominal pain per week
need for interventional laxative | 1 week
  need for rescue treatment (osmotic laxative: lactulose 1 ml of syrup per 1 kg of body weight) when no stool passed for 3 consecutive days)
flatulence | 1 week
  number of episodes of flatulence per 1 week
adverse events | 4 weeks
  any adverse events (mild or seriuos) reported by parents during the study period(pain, infections, hospitalizations, accidents or any other event related or not related to study intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Hania Szajewska, Professor, Study Director — The Medical University of Warsaw
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw, Poland

REFERENCES:
- [Background] Hyman PE, Milla PJ, Benninga MA, Davidson GP, Fleisher DF, Taminiau J. Childhood functional gastrointestinal disorders: neonate/toddler. Gastroenterology. 2006 Apr;130(5):1519-26. doi: 10.1053/j.gastro.2005.11.065. PMID 16678565
- [Result] Belsey J, Greenfield S, Candy D, Geraint M. Systematic review: impact of constipation on quality of life in adults and children. Aliment Pharmacol Ther. 2010 May;31(9):938-49. doi: 10.1111/j.1365-2036.2010.04273.x. Epub 2010 Feb 20. PMID 20180788
- [Result] Pijpers MA, Tabbers MM, Benninga MA, Berger MY. Currently recommended treatments of childhood constipation are not evidence based: a systematic literature review on the effect of laxative treatment and dietary measures. Arch Dis Child. 2009 Feb;94(2):117-31. doi: 10.1136/adc.2007.127233. Epub 2008 Aug 19. PMID 18713795
- [Result] Loening-Baucke V, Miele E, Staiano A. Fiber (glucomannan) is beneficial in the treatment of childhood constipation. Pediatrics. 2004 Mar;113(3 Pt 1):e259-64. doi: 10.1542/peds.113.3.e259. PMID 14993586
- [Result] Staiano A, Simeone D, Del Giudice E, Miele E, Tozzi A, Toraldo C. Effect of the dietary fiber glucomannan on chronic constipation in neurologically impaired children. J Pediatr. 2000 Jan;136(1):41-5. doi: 10.1016/s0022-3476(00)90047-7. PMID 10636972
- [Derived] Chmielewska A, Horvath A, Dziechciarz P, Szajewska H. Glucomannan is not effective for the treatment of functional constipation in children: a double-blind, placebo-controlled, randomized trial. Clin Nutr. 2011 Aug;30(4):462-8. doi: 10.1016/j.clnu.2011.01.012. Epub 2011 Feb 12. PMID 21320737